CLINICAL TRIAL: NCT01444872
Title: A Randomized, Single-Blind, Placebo-Controlled, Adaptive, Ascending Dose Study to Evaluate the Effects of TRV120027 on Renal Pharmacodynamics in Patients With Heart Failure and Mild to Moderate Renal Dysfunction
Brief Title: Study to Evaluate TRV120027 on Renal Pharmacodynamics in Patients With Heart Failure and Renal Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trevena Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: CP120027.1002
Record Dates: First submitted 2011-09-19; First posted 2011-10-03 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-08

CONDITIONS: Heart Failure; Kidney Disease
MeSH Terms: conditions — Heart Failure; Kidney Diseases | interventions — Sar-Arg-Val-Tyr-Ile-His-Pro-Ala-OH; Saline Solution

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- TRV120027 (Experimental): TRV120027 administered as an IV infusion
  Interventions: Drug: TRV120027
- Normal Saline (Placebo Comparator): Normal Saline administered as an IV infusion
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: TRV120027 — IV infusion
  Arms: TRV120027
Drug: Normal Saline — IV infusion
  Arms: Normal Saline

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of TRV120027 in subjects with heart failure and mild to moderate renal dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent
* Heart Failure
* Mild to moderate renal dysfunction
* Age 18- <75
* Males and females (non-childbearing potential)

Exclusion Criteria:

* Any significant disease or condition that would interfere with the interpretation of safety or efficacy or efficacy data as determined by the Investigator based on medical history, physical examination or laboratory tests
* Any other serious life threatening disease that may impair the interpretation of safety or efficacy data from the study as determined by the Investigator
* Allergy or clinically-significant intolerance to ARBs or ACE inhibitors
* Clinical signs or symptoms of acute decompensated heart failure
* Pregnant or lactating

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-08; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Glomerular Filtration Rate | Every hour during final 6 hours of study drug infusion
  Assessments of glomerular filtration rate are made hourly during the 6-hour study drug infusion on study Day 1 and study Day 3. GFR in hours 4-6 are compared to GFR in hours 1-3, and comparisons made between Placebo and TRV120027.
Change from Baseline in Vital Signs (Blood pressure, heart rate) | Baseline, during infusion, and following infusion, on Study Day 1 and Study Day 3
  Vital signs measurements made during and following drug infusion will be evaluated as a change from baseline, and comparing placebo to TRV120027. Assessments are made on study Day 1 and study Day 3.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Orlando Clinical Research Center, Orlando, Florida
  - DaVita Clinical Research, Minneapolis, Minnesota
  - Duke Clinical Research Unit, Durham, North Carolina
  - New Orleans Center for Clinical Research, Knoxville, Tennessee

REFERENCES:
- See also: Sponsor's Website — http://www.trevenainc.com